CLINICAL TRIAL: NCT06478303
Title: LAnguage-Motor Imagery Circuits to Improve Motor Learning and Language Comprehension
Acronym: LAMI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University of Burgundy (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0349; 2023-A02322-43 (Other: ID RCB)
Record Dates: First submitted 2024-06-13; First posted 2024-06-27 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Corticospinal Excitability; Cortical Activation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- TMS Experimental group
  Interventions: Other: Motor imagery; Other: Action reading
- fMRI Experimental group
  Interventions: Other: Motor imagery; Other: Action reading; Other: Motor localizer
- Experimental ccPAS group
  Interventions: Other: Motor imagery; Other: Action reading
- Sham ccPAS group
  Interventions: Other: Motor imagery; Other: Action reading
- control group
  Interventions: Other: Motor imagery; Other: Action reading

INTERVENTIONS:
Other: Motor imagery — Participants were asked to imagine arm or foot movements.
Other: Action reading — Participants were asked to read sentences involving arm or foot movements
Other: Motor localizer — Participants were asked to perform arm or foot movements
  Groups: fMRI Experimental group

SUMMARY:
Recent evidence suggests that cognitive systems do not operate in isolation but interact within broader networks, thus opening new avenues for fundamental and clinical research. An illustrative example is the interaction between language comprehension and motor representations. For instance, motor training (e.g., sports, origami training) can facilitate action verb recognition, whereas motor deficits (e.g., upper limb immobilization) can hinder the processing of action language. Similarly, action language has been shown to affect motor performance. These effects are attributed to an implicit form of motor imagery, an automatic simulation of motor experience (without actual movement) evoked by action words. Interestingly, literature supports the idea that the motor simulations used for imagining an action are also engaged during the reading of action language, leading to similar neurophysiological and behavioral changes in both processes. However, questions remain about the similarity of the simulations generated by motor imagery and action language. This project, encompassing three experimental sequences, aims to address these questions to achieve significant scientific advancements in both theoretical and applied domains.

ELIGIBILITY:
Inclusion Criteria:

* persons who have given written consent,
* healthy subjects
* subjects reading and understanding French
* right-handed,
* affiliated with a social security system,
* between 18 and 40 years old,
* had completed the TMS inclusion questionnaire or had undergone a medical examination prior to participation in the MRI study.

Exclusion Criteria:

* Existence of a severe general medical condition: cardiac, respiratory, hematological, renal, hepatic, cancerous,
* Regular use of anxiolytics, sedatives, antidepressants, neuroleptics,
* Characterized psychiatric pathology,
* Ingestion of alcohol prior to the examination,
* Persons covered by articles L1121-5 to L1121-8 of the CSP,
* Presence of contraindications to MRI or TMS.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be aged between 18 and 40, reading and understanding French, with no neurological or psychiatric disorders, no uncorrected vision deficits, and meeting all MRI or TMS examination criteria. they were recruited at the University of Burgundy (TMS measures only) and the University of Grenoble Alpes (fMRI measures only).
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2024-07-27 (Actual); Primary Completion 2027-07-26 (Estimated); Study Completion 2028-07-26 (Estimated)

PRIMARY OUTCOMES:
Level of corticospinal excitability | 1 hour and 30 minutes
  this is a physiological response obtained by transcranial magnetic pulses (TMS). This is an indicator of the excitability of the motor system, which can be used at rest or during various cognitive tasks (motor imagery or action reading).
Cortical activation (BOLD signal) | 1 hour
  this is a cortical response obtained via a fMRI. This is an indicator of the brain activity, which can be used at rest or during motor and cognitive tasks (motor imagery or action reading).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent VERCUEIL, Principal Investigator — CHU Grenoble Alpes
Locations (2):
- France (2):
  - CHU Grenoble Alpes, Grenoble, Grenob
  - Université de Bourgogne, Dijon